CLINICAL TRIAL: NCT03236259
Title: The Effect of Berry Extract Administration on Cognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: BioActor B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Brainport-001
Record Dates: First submitted 2017-07-20; First posted 2017-08-01 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Impairment; Overweight and Obesity
MeSH Terms: conditions — Cognitive Dysfunction; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brainport high dose (Active Comparator)
  Interventions: Dietary Supplement: Brainport high dose
- Brainport low dose (Active Comparator)
  Interventions: Dietary Supplement: Brainport low dose
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Brainport high dose — berry extract, high dose. Daily ingestion of capsule
  Arms: Brainport high dose
Dietary Supplement: Brainport low dose — Berry extract, low dose. Daily ingestion of capsule
  Arms: Brainport low dose
Dietary Supplement: Placebo — Maltodextrin. Daily ingestion of capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of daily supplementation of Brainport for a period of 6 months on cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* Age between 40 and 60 years
* BMI 25 - 35 kg/m2

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat). Dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and /or laboratory assessments that might limit participation in or completion of the study protocol.
* Diabetes
* Use of medication that might have influence on endpoints (hypertension medication)
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study in the 180 days prior to the study
* Use of antibiotics in the 30 days prior to the start of the study
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Pregnancy, lactation
* Abuse of products (> 20 alcoholic consumptions per week and drugs)
* Smoking
* Weight gain or loss (> 3 kg in previous 3 months)
* High physical activity (>4.5 hours of running/week)
* History of any side effects towards intake of berries

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Cognition | 6 months
  test attention with STROOP
Cognition | 6 months
  Test concentration with 'cijferdoorstreep test'
Cognition | 6 months
  Test psychomotor speed with grooved pegboard

SECONDARY OUTCOMES:
vascular structure | 6 months
  measure vascular structure with ultrasound.
Mood | 6 months
  Test mood with visual analogue mood scale. 8 emotions are scored on a 1-10 scale.
Blood pressure | 6 months
Liver function | 6 months
  analysis of alkaline phosphatase, alanine aminotransferase, aspartaat aminotransferase, bilirubine, gamma-glutamyltransferase to determine liver function.
flavo-enzyme | 6 months
  monoamine oxidase B analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands